CLINICAL TRIAL: NCT07393633
Title: Assessing Whole-body Metabolism in Gynecologic Cancers in Response to a Single Chemotherapy Cycle and/ or Immunotherapy
Status: Completed | Type: Observational
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 5204
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Cancers
Keywords: gynecologic cancer; whole body metabolism; lipid metabolism; ovarian cancer; cardiometabolic outcomes; uterine cancer; resting metabolic rate; oxygen consumption; carbon dioxide production
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with biopsy proven gynecologic cancer: Patients with biopsy proven gynecologic cancer undergoing active treatment

SUMMARY:
It is well established that cancer cells have fundamentally altered metabolism, which contributes to tumorigenicity and malignancy. For years, research findings supported that the universal property of all cancer cells was to increase glycolytic flux for anaerobic glycolysis (i.e., Warburg effect), which was accepted as the dominant pathway for energy metabolism. Fortunately, by understanding these changes in cellular metabolism multiple new approaches to cancer therapy, focused on reprogramming the energy metabolism of the cell. Recently, further investigation in the field found that cancer cells exhibit multiple alterations in metabolic pathways, not only glycolysis.

Alterations in lipid metabolism in cancer cells have recently been recognized as potential targets for therapeutic interventions due to its role in cellular proliferation, energy storage, and the generation of signaling molecules. Numerous cancer types can rely on lipids as an energy source, increasing fatty acid synthesis and degradation to promote proliferation and metastasis. Several therapeutic agents utilized in gynecologic malignancies impact lipid metabolism.

The objective of the proposed study will be to determine the impact of cancer directed therapy on the lipid metabolism of non-malignant tissues. No study to date has assessed whole-body lipid metabolism in patients undergoing chemotherapy (i.e. cytotoxic chemotherapy and/or immunotherapy). These novel findings will provide crucial knowledge about the dysregulation of whole-body metabolism in patients receiving chemotherapy for treatment of gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age >18 years
* Biopsy confirmed gynecologic cancer.
* Scheduled to or currently undergoing infusion therapy.
* Receiving cytotoxic chemotherapy or immunotherapy.

Exclusion Criteria:

* Inability to provide voluntary informed consent.
* Received inpatient medical intervention for adverse effects of chemotherapy.
* Circumstances and/or medical condition that would limit compliance with study requirements and protocol, as determined by the principal investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecologic cancer engaged in active treatment.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2026-01-24 (Actual)

PRIMARY OUTCOMES:
Fasting Whole Body Carbon Dioxide Production - Baseline | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting whole body carbon dioxide production (VCO2), which is assessed using indirect calorimetry and measured in ml/min.
Fasting Whole Body Oxygen Consumption - Baseline | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting whole body oxygen consumption (VO2), which is assessed using indirect calorimetry in ml/min
Fasting Resting Metabolic Rate (RMR) - Baseline | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting resting metabolic rate (RMR), which is assessed using indirect calorimetry and measured in kcal/day.
Fasting respiratory exchange ratio (RER) - Baseline | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting respiratory exchange ratio (RER), which is assessed using indirect calorimetry.
Fasting Whole Body Carbon Dioxide Production - 30 Minutes Post | Fasting, measured 30 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting whole body carbon dioxide production (VCO2), which is assessed using indirect calorimetry and measured in ml/min.
Fasting Whole Body Oxygen Consumption - 30 Minutes Post | Fasting, measured 30 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting whole body oxygen consumption (VO2), which is assessed using indirect calorimetry in ml/min
Fasting Resting Metabolic Rate (RMR) - 30 Minutes Post | Fasting, measured 30 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting resting metabolic rate (RMR), which is assessed using indirect calorimetry and measured in kcal/day.
Fasting respiratory exchange ratio (RER) - 30 Minutes Post | Fasting, measured 30 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting respiratory exchange ratio (RER), which is assessed using indirect calorimetry.
Fasting Whole Body Carbon Dioxide Production - 90 Minutes Post | Fasting, measured 90 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting whole body carbon dioxide production (VCO2), which is assessed using indirect calorimetry and measured in ml/min.
Fasting Whole Body Oxygen Consumption - 90 Minutes Post | Fasting, measured 90 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting whole body oxygen consumption (VO2), which is assessed using indirect calorimetry in ml/min
Fasting Resting Metabolic Rate (RMR) - 90 Minutes Post | Fasting, measured 90 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting resting metabolic rate (RMR), which is assessed using indirect calorimetry and measured in kcal/day.
Fasting respiratory exchange ratio (RER) - 90 Minutes Post | Fasting, measured 90 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting respiratory exchange ratio (RER), which is assessed using indirect calorimetry.
Fasting Whole Body Carbon Dioxide Production - 150 Minutes Post | Fasting, measured 150 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting whole body carbon dioxide production (VCO2), which is assessed using indirect calorimetry and measured in ml/min.
Fasting Whole Body Oxygen Consumption - 150 Minutes Post | Fasting, measured 150 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting whole body oxygen consumption (VO2), which is assessed using indirect calorimetry in ml/min
Fasting Resting Metabolic Rate (RMR) - 150 Minutes Post | Fasting, measured 150 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting resting metabolic rate (RMR), which is assessed using indirect calorimetry and measured in kcal/day.
Fasting respiratory exchange ratio (RER) - 150 Minutes Post | Fasting, measured 150 minutes after the start of a single cancer treatment during the study visit at one time point during active cancer treatment.
  Fasting respiratory exchange ratio (RER), which is assessed using indirect calorimetry.

SECONDARY OUTCOMES:
Fasting capillary blood glucose | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting capillary blood glucose (mg/dL)
Fasting capillary blood lactate | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting capillary blood lactate (mmol/L)
Fasting venous blood glucose | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous plasma glucose (mg/dL)
Fasting venous blood insulin | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous serum insulin (µlU/mL)
Fasting venous blood lactate | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous plasma blood lactate (mmol/L)
Fasting venous cholesterol (mg/dL) | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous cholesterol (mg/dL)
Fasting venous HDL (mg/dL) | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous HDL (mg/dL)
Fasting venous LDL (mg/dL) | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous LDL (mg/dL)
Fasting venous VLDL (mg/dL) | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous VLDL (mg/dL)
Fasting venous triglycerides (mg/dL) | Fasting, measured at the start of the study visit at one time point during active cancer treatment.
  Fasting venous triglycerides (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets will not be publicly available but can be shared by request.
Supporting Information: Study Protocol